CLINICAL TRIAL: NCT03738904
Title: Prospective Randomized Controlled Trial of an Enhanced Recovery Protocol for Anorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00054080
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Anorectal Disorder
MeSH Terms: conditions — Rectal Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (multimodal ERAS) (Experimental): Arm1 (Multimodal ERAS):
  Preoperative:
  oral gabapentin 600mg and oral acetaminophen 1,000mg
  Postoperative pain control:
  1. Gabapentin oral 300 mg TID (#42, refill #1)
  2. Acetaminophen oral 1000mg TID (#42, refill #1)
  3. Ketorolac oral 10 mg TID (#15, refill #0)
  4. Oxycodone oral 5 mg PRN every 6 hours (#30, refill #0)
  Postoperative laxative regimen:
  1. Daily MiraLAX 1 scoop in 1 glass of water for 15 days
  2. Daily milk of magnesia 1 tablespoon if no bowel movement by POD2 until regular bowel movements
  3. Daily mineral oil 1 table spoon if no bowel movement by POD2 until regular bowel movements
  Interventions: Combination Product: ERAS
- Arm 2 (control) (Active Comparator): Postoperative pain control:
  1. Oxycodone oral 5 mg PRN every 6 hours (#30, refill #0)
  2. Patients will be allowed to take oral acetaminophen and ibuprofen over the counter if needed but active narcotic-sparing pain management regimen will not be implemented
  Postoperative laxative regimen:
  1. Daily MiraLAX 1 scoop in 1 glass of water for 15 days
  2. Daily milk of magnesia 1 tablespoon if no bowel movement by POD2 until regular bowel movements Daily mineral oil 1 table spoon if no bowel movement by POD2 until regu-lar bowel movements
  Interventions: Combination Product: Standard of care

INTERVENTIONS:
Combination Product: ERAS — Gabapentin Acetaminophen Ketoroloac IV (intraop) and PO Dexamethasone (included with benzocaine in local anesthesia) Oxycodone PO Polyethylene glycol
  Arms: Arm 1 (multimodal ERAS)
Combination Product: Standard of care — Oxcodone PO Ketorolac IV only (intraop)
  Arms: Arm 2 (control)

SUMMARY:
The purpose of the study is to evaluate whether being randomized to an aggressive postoperative non-narcotic pain regimen that treats pain from multiple different pathways may decrease postoperative pain levels, decrease constipation, and decrease the dependency on opioid medications after anorectal surgery versus the standard of care for managing pain. This use of a more aggressive pain regimen is considered an enhanced recovery after surgery (ERAS) protocol because it is theorized to improve or "enhance" postoperative recovery by both decreasing the use of narcotics and their detrimental effects as well as increasing the benefit of using additional non-narcotic pain medication.

DETAILED DESCRIPTION:
Although pain is a predictable part of the postoperative experience, inadequate management of pain is common and can have profound implications Most patients who undergo surgical procedures experience acute postoperative pain, but evidence suggests that less than half report adequate postoperative pain relief. Many preoperative, intraoperative, and postoperative interventions and management strategies are available for reducing and managing postoperative pain. Mostly, pain is treated with opioids which are narcotics. medically they are primarily used for pain relief and these are historically considered "safe" drugs as they do not impose an increased risk of bleeding, kidney, or stomach problems. However, many patients taking high dose opioids have a higher risk of constipation. Unrelieved postoperative pain may result in economic and medical implications such as extended lengths of stay, readmissions, and patient dissatisfaction with medical care. With the rising concern over narcotic use, physicians are increasingly seeking alternative ways to help patients manage pain throughout their hospital stay and beyond However, few studies in anorectal surgery have shown that using an aggressive postoperative non-narcotic pain regimen (ERAS) can help reduce postoperative pain and decreased returns to emergency care.

ELIGIBILITY:
Inclusion Criteria:

* Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
* Males or females, age 18 to 70 years old at the time of study screening;
* American Society of Anesthesiologists (ASA) Class I-III (Appendix III) undergoing elective anorectal surgery
* Patients undergoing the following hemorrhoid surgeries will be included:
* Excisional single column or multiple column hemorrhoidectomy including internal and external component
* Stapled hemorrhoidpexy (aka procedure for prolapsed hemorrhoids with or without excision of external hemorrhoid or skin tag)
* Trans anal hemorrhoidal dearterialization with mucopexy (THD) with or without excision of external hemorrhoid or skin tag
* Patients undergoing the following anal fistula surgery will be included:
* Anal fistulotomy or fistulectomy of intersphincteric or tran-sphincteric fistula with wound > 1 cm
* Endorectal or an cutaneous advancement flap for anal fistula re-pair

Exclusion Criteria:

* Unable or unwilling to provide informed consent or comply with study procedures
* American Society of Anesthesiologists (ASA) Class IV or V; emergency surgeries
* Children <18
* Patients over age 70 due to small risk of altered mental status with gabapentin in elderly6
* Patients with impaired renal clearance (baseline creatinine 1.5mg/dL, creatinine clearance < 60ml/min or known renal dysfunction)
* Patients with known liver dysfunction (Childs class A, B, or C)
* Patients with prior liver or kidney transplant
* Pregnant patients
* Patients requiring emergency surgery
* Patients taking narcotics or steroids at the time of surgery
* Patients having external hemorrhoidectomy or skin anal tag excision only
* Patients having anal abscess drainage, seton placement without definitive fistula repair, or ligation of intersphincteric fistula tract, subcutaneous fistulotomy or fistulotomy with wound <1 cm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao LY, Parrish AB, Fleshner PR, Zaghiyan KN. Implementation of a Multimodal Enhanced Recovery Protocol in Ambulatory Anorectal Surgery: A Randomized Trial. Dis Colon Rectum. 2024 Oct 1;67(10):1304-1312. doi: 10.1097/DCR.0000000000003435. Epub 2024 Jul 17. PMID 39016381

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Multimodal ERAS): Arm1 (Multimodal ERAS):
  Preoperative:
  oral gabapentin 600mg and oral acetaminophen 1,000mg
  Postoperative pain control:
  1. Gabapentin oral 300 mg TID (#42, refill #1)
  2. Acetaminophen oral 1000mg TID (#42, refill #1)
  3. Ketorolac oral 10 mg TID (#15, refill #0)
  4. Oxycodone oral 5 mg PRN every 6 hours (#30, refill #0)
  Postoperative laxative regimen:
  1. Daily MiraLAX 1 scoop in 1 glass of water for 15 days
  2. Daily milk of magnesia 1 tablespoon if no bowel movement by POD2 until regular bowel movements
  3. Daily mineral oil 1 table spoon if no bowel movement by POD2 until regular bowel movements
  ERAS: Gabapentin Acetaminophen Ketoroloac IV (intraop) and PO Dexamethasone (included with benzocaine in local anesthesia) Oxycodone PO Polyethylene glycol
- Arm 2 (Control): Postoperative pain control:
  1. Oxycodone oral 5 mg PRN every 6 hours (#30, refill #0)
  2. Patients will be allowed to take oral acetaminophen and ibuprofen over the counter if needed but active narcotic-sparing pain management regimen will not be implemented
  Postoperative laxative regimen:
  1. Daily MiraLAX 1 scoop in 1 glass of water for 15 days
  2. Daily milk of magnesia 1 tablespoon if no bowel movement by POD2 until regular bowel movements Daily mineral oil 1 table spoon if no bowel movement by POD2 until regu-lar bowel movements
  Standard of care: Oxcodone PO Ketorolac IV only (intraop)
Period: Overall Study
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control)
Started | 54 | 55
Completed | 45 | 44
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control) | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 38 [20 to 67] | 38 [23 to 59] | 38 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 20 | 28 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Use Postoperatively in Oral Morphine Equivalents
Description: Total amount of narcotics used
Time Frame: 1 week postoperatively
Measure: Median (Full Range); unit: Oral morphine miligram equivalents
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control)
Number analyzed (Participants) | 45 | 44
Oral morphine miligram equivalents | 8 [0 to 390] | 79 [0 to 600]

2. Secondary Outcome: Median Postoperative Pain Scores
Description: Level of pain measured on a scale of 0-10 with 0 being the lowest level of pain and 10 being the highest level of pain as reported by the participant
Time Frame: 1 week postoperatively
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control)
Number analyzed (Participants) | 45 | 44
score on a scale | 4 [0 to 10] | 6 [0 to 10]

3. Secondary Outcome: Complications
Description: Number of participants who experienced complications
Time Frame: 1 month postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control)
Number analyzed (Participants) | 45 | 44
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Description: Any unexpected or adverse event that may or may not have resulted in unplanned visit to the emergency department, clinic, or additional tests or procedures.
Arm/Group | Arm 1 (Multimodal ERAS) | Arm 2 (Control)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 4/45 | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Multimodal ERAS) (N=45) | Arm 2 (Control) (N=44)
Adverse event not resulting in significant morbidity or mortality (Surgical and medical procedures) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03738904/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT03738904/ICF_001.pdf